CLINICAL TRIAL: NCT06988540
Title: Evaluation of a Telehealth Personal Health Planning Program for Patients With Uncontrolled Type 2 Diabetes
Brief Title: T2D Pilot Study for Patients With Uncontrolled Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00110685
Record Dates: First submitted 2025-05-16; First posted 2025-05-25 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-04

CONDITIONS: Diabetes Mellitus; Health Behavior; Diabetes Mellitus, Type 2; Group Meetings
MeSH Terms: conditions — Diabetes Mellitus; Health Behavior; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with intervention receiving a 16 week personalized health plan and control group receiving usual care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Health Planning Program Participant with Type 2 Diabetes (Experimental): A novel virtual group visit care model for individuals with T2D for long-term health improvements and disease management. This intervention group will receive a 16-week virtual, Personal Health Planning (PHP) T2D Program emphasizing behavioral engagement, utilizing a mixed methods research design. Outcomes include cardiometabolic labs and surveys.
  Interventions: Other: Personalized Health Planning Program Administration
- Usual Care (Type 2 DM) (Placebo Comparator): The control group will receive usual care. They will be asked to have laboratory tests and answer survey questions regarding diabetes distress and diabetes empowerment.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Personalized Health Planning Program Administration — The T2D PHP program is 8 hour-long sessions offered over 16 weeks. The program includes development of a personal health plan supported by a patient-provider health risk assessment; group session structure supplemented by educational, video sessions; lessons, discussions, and activities based on behavioral modification, health engagement, and diabetes distress; goal progress tracking; social support; mindful awareness practices and qualitative health evaluations via surveys and a one-on-one consultation with a personal health coach. Participants will be provided a group participant notebook that provides information discussed during the program. The T2D PHP program is a complement to routine care.
  Arms: Personalized Health Planning Program Participant with Type 2 Diabetes
Other: Usual Care — Patients will be encouraged to see their diabetes provider. Patients will not participate in the T2D PHP program but will complete laboratory tests and surveys as listed in the section on outcomes.
  Arms: Usual Care (Type 2 DM)

SUMMARY:
The primary objective of the study is to evaluate implementation and determine the effectiveness of a telehealth personal health planning program for individuals with uncontrolled Type 2 Diabetes Mellitus. For this study, participants will be randomized into either the Telehealth Program or the standard of care group. The personal health planning (PHP) Type 2 Diabetes program is a virtual, 8 session/16- week behavioral health program. The program includes development of a personal health plan supported by a patient-provider health risk assessment; group session structure supplemented by educational, on-demand video sessions; lessons, discussions, and activities based on understanding behavioral modification, health engagement, and diabetes distress; goal progress tracking; social support; mindful awareness practices; 3 and 6-month post program sessions and qualitative health evaluations via surveys and a one-on-one consultation with a personal health coach. Those in the control group will receive usual care by the participants personal care team. All participants will come to the Duke Research at Pickett Road facility for a pre and post-program fasting A1C and lipid panel blood draw (if required).

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes diagnosis
* 18 and over
* 2 A1C results in last 18 months
* A1C of 8-12
* Access to a electronic device with internet
* Duke Patient

Exclusion Criteria:

* Type 1 Diabetes
* Pregnant
* Blind
* Deaf
* Cognitive Impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Day 1 (Preintervention) and Month 5 (Postintervention)
  Blood test to determine average blood sugar

SECONDARY OUTCOMES:
Attendance at Personalized Health Program Group Meetings | 16 weeks
Diabetes Empowerment Scale | Day 1 (Preintervention) and Month 5 (Postintervention)
  The Diabetes Empowerment Scale (DES) is a tool designed to measure the psychosocial self-efficacy of people with diabetes. It helps assess how confident individuals feel about managing their diabetes and making necessary lifestyle changes. The DES consists of 28 items divided into three subscales: Managing the Psychosocial Aspects of Diabetes, Assessing Dissatisfaction and Readiness to Change, Setting and Achieving Goals. Each item on the DES is rated on a 5-point Likert scale, with 1 indicating strongly disagree and 5 indicating strongly agree. Total score is obtained by dividing by number of questions answered so total score range would be 1-5. Higher scores indicate greater empowerment and confidence in managing diabetes. Lower scores suggest areas where the individual may need more support or education
Diabetes Distress | Day 1 (Preintervention) and Month 5 (Postintervention)
  The Diabetes Distress Scale (DDS) is a tool designed to measure the emotional burden and stress associated with managing diabetes. It consists of 17 items that assess various aspects of diabetes-related distress over the past month 1. Each item, subdomain scale, and total scale is rated on a 6-point scale, ranging from 1 (not a problem) to 6 (a very serious problem). The subdomains are: Emotional Burden Physician-related Distress Regimen-related Distress Interpersonal Distress
Triglycerides | Day 1 (Preintervention) and Month 5 (Postintervention)
  Triglycerides is a type of lipid measurement
HDL Cholesterol | Day 1 (Preintervention) and Month 5 (Postintervention)
  HDL Cholesterol is a type of lipid measurement
LDL Cholesterol | Day 1 (Preintervention) and Month 5 (Postintervention)
  LDL Cholesterol is a type of lipid measurement
Total Cholesterol | Day 1 (Preintervention) and Month 5 (Postintervention)
  Total Cholesterol is a type of lipid measurement
Body Mass Index (BMI) | Day 1 (Preintervention) and Month 5 (Postintervention)
  A measure of weight standardize for height to assess whether patient is considered normal, overweight, or obese
Systolic Blood Pressure | Day 1 (Preintervention) and Month 5 (Postintervention)
Diastolic Blood Pressure | Day 1 (Preintervention) and Month 5 (Postintervention)
Hemoglobin A1c | Month 17
  Blood test to determine average blood sugar
Patient Goals Progress | Sessions 3-8 during the intervention
  Participant rated success based on a 1-5 likert scale, 5 being higher success rate
Fasting Plasma Glucose | Day1 (preintervention), Month 5 (post intervention), Month 17 (1 year post intervention)

OTHER OUTCOMES:
Diabetes Care Profile | Day 1 (preintervention)
  The DCP is a self-administered questionnaire that assesses the social and psychological factors related to diabetes and its treatment. The instrument contains 234 items and sixteen scales. These scales assess diabetes attitudes, diabetes beliefs, self-reported diabetes self-care, and difficulties with diabetes mgt. IT will be administered pre intervention to personalize each individual's care plan.
Post Program Satisfaction | Month 5 (Postintervention)
  Post Program Satisfaction for intervention group only
Patient Goals | Obtained during sessions 3-8 during the intervention for the intervention group
  Patient selected diabetes management goals

CONTACTS AND LOCATIONS:
Overall Officials: Susan E Spratt, MD, Principal Investigator — Duke University
Locations (1):
- Duke Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No